CLINICAL TRIAL: NCT01631695
Title: Evaluation of the Performances of Medasense Pain Monitor During General Anesthesia and Postoperative Recovery Compared to Pain Related Physiological Indicators and to Subjective Assessment of Pain by Anesthesiologist
Brief Title: Clinical Evaluation of Medasense Pain Monitor Performances
Status: Completed | Type: Observational
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: Medasense002; 0281-09-RMB (Other: Rambam Health Care Campus, Haifa, Israel)
Record Dates: First submitted 2011-10-24; First posted 2012-06-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Surgery; Pain; Postoperative Pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the performances of Medasense's non-invasive pain monitoring is compared with standard pain related indicators, such as heart rate, galvanic skin response, etc. , and with a subjective pain level assessment. The subjective pain level is assessed by the anesthesiologist when the patient is under general anesthesia and by the patient and a nurse in post anesthetic care unit (PACU).

The study is based on recording and analyzing the subject's physiological signals, while recording painful events, medication dosing and different clinical signs.

DETAILED DESCRIPTION:
Pain is an unpleasant sensation, ranging from slight discomfort to intense suffering. Since pain is a subjective phenomenon, it has frequently defied objective, quantitative measurements. Today, in order to measure pain, subjective uni-dimensional scales are used to quantify pain. One of the most common scale used to rate a patient's pain intensity is the visual analog scale (VAS), usually scored from 0 to 100. Hitherto, those scales are based on the subjective evaluation of pain by the patient.

During anesthesia the patient cannot communicate and therefore the verbal or other report is impossible. Therefore, due to misrepresentation of the existence or extent of pain, care providers may fail to estimate the correct measure of pain and give too much or too little medication. A scoring system of pain level is therefore needed. That is the problem Medasense's system tries to approach.

In this study investigators intend to test and analyze the performances of Medasense pain monitor by comparing its results with standard pain related indicators and with subjective patient's pain level assessment. The patient's pain level will be assessed by the anesthesiologist during surgery based on known pain stimuli, medications administered and clinical signs, and by the PACU nurse and patient's reports, when the patient is in recovery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2
* Elective surgery under general anesthesia
* Baseline blood pressure < (170\100 mmHg), heart rate < 100 bpm

Exclusion Criteria:

* Pregnancy or lactation
* History of severe cardiac arrhythmias
* Presence of any neuromuscular or neurological disease
* Use of central nervous system (CNS) -active medications
* Abuse of alcohol or illicit drugs
* History of mental retardation or any mental disease
* Any severe lung, liver, renal disease and uncontrolled diabetes mellitus
* Use of a α or β-adrenergic antagonist or anticholinergics
* Allergy to any of the drugs to be used during surgery
* Use of regional anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgeries under general anesthesia, healthy or suffering from minor chronic diseases (ASA I-II)
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in Medasense's non-invasive pain monitoring index in response to painful events. | before versus after painful stimuli (for instance: intubation, skin incision, trocar insertion)
  outcome measure will be assessed one minute before painful event, and will be compared to a measure taken during the painful event.

SECONDARY OUTCOMES:
Changes in all pain related physiological parameters (heart rate, heart rate variability, Plethysmograph amplitude, skin conductance, etc) in response to specific painful stimuli | before versus after painful stimuli (for instance: intubation, skin incision, trocar insertion)
  Outcome measures will be assessed one minute before painful event, and will be compared to measures taken during the painful event.
Changes in anesthesiologist subjective pain assessment in response to specific painful stimuli | before versus after painful stimuli (for instance: intubation, skin incision, trocar insertion)
  Outcome measure will be assessed one minute before painful event, and will be compared to a measure taken during the painful event.
Changes in Medasense index/pain related parameters/subjective pain assessment in response to changes in the level of analgesic drugs | before versus after analgesic drug administration
  Outcome measures will be assessed one minute before administration of analgesic drug, and will be compared to measures taken one minute after.
  Participants will be followed for the duration of surgery and Postoperative Recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Edry, MD, Principal Investigator — Department of Anesthesiology, Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Treister R, Kliger M, Zuckerman G, Aryeh IG, Eisenberg E. Differentiating between heat pain intensities: the combined effect of multiple autonomic parameters. Pain. 2012 Sep;153(9):1807-1814. doi: 10.1016/j.pain.2012.04.008. Epub 2012 May 29. PMID 22647429
- [Result] Ben-Israel N, Kliger M, Zuckerman G, Katz Y, Edry R. Monitoring the nociception level: a multi-parameter approach. J Clin Monit Comput. 2013 Dec;27(6):659-68. doi: 10.1007/s10877-013-9487-9. Epub 2013 Jul 9. PMID 23835792